CLINICAL TRIAL: NCT03886623
Title: A Systematic Oral Care Program in Post-Mechanically Ventilated, Post-Intensive Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Esther Chipps, Director HS Nursing Quality & Research, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011H0015
Record Dates: First submitted 2012-10-09; First posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Methicillin-resistant Staphylococcus Aureus; Methicillin-Sensitive Staphylococcus Aureus Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4-day systematic oral hygiene (Experimental): The intervention proposed would include a 4-5 day systematic oral hygiene program. Using a pea-sized amount of Colgate Total Clean Mint Toothpaste with a Battery-operated Oral-B Pro-Health Type 3744 toothbrush, all surfaces, tongue-side, check-side, and biting surfaces of the participants teeth will be brushed. The tongue will be brushed with a GUM Dual Action Tongue Cleaner and flossing will be done with GUM Flossmate handle and Oral B Guide Floss in between the contacts of each tooth. The mouth will then be rinsed with Crest Pro-Health mouthwash rinse for 30 seconds twice daily. A Medline Remedy Phytoplex lip balm will then be applied.
  Interventions: Procedure: 4-day systematic oral hygiene
- Standard of Care oral care (Other): Standard of Care oral care. Currently, the intensive care units utilize a commercially available pre-package oral hygiene kit. This includes mouthwash swabbing every 2 hours with Careline Alcohol-Free mouthwash or Sage Alcohol Free mouthwash, teeth brushing (with Sage Toothette Oral Care, Sodium Bicarbonate Toothpaste and Sage Suction Toothbrush) every 12 hours, deep oral suctioning every 8 hours and prior to oral Endotracheal tube (ET) retaping, and Paroex Oral Rinse chlorohexidine gluconate (15ml) swabbed onto oral surfaces every 12 hours (SICU patients only). Mouth care is documented every two hours.
  Interventions: Other: Standard of Care oral care

INTERVENTIONS:
Procedure: 4-day systematic oral hygiene — he intervention proposed would include a 4-5 day systematic oral hygiene program. Using a pea-sized amount of Colgate Total Clean Mint Toothpaste with a Battery-operated Oral-B Pro-Health Type 3744 toothbrush, all surfaces, tongue-side, check-side, and biting surfaces of the participants teeth will be brushed. The tongue will be brushed with a GUM Dual Action Tongue Cleaner and flossing will be done with GUM Flossmate handle and Oral B Guide Floss in between the contacts of each tooth. The mouth will then be rinsed with Crest Pro-Health mouthwash rinse for 30 seconds twice daily. A Medline Remedy Phytoplex lip balm will then be applied.
  Arms: 4-day systematic oral hygiene
Other: Standard of Care oral care — Standard of Care oral care. Currently, the intensive care units utilize a commercially available pre-package oral hygiene kit. This includes mouthwash swabbing every 2 hours with Careline Alcohol-Free mouthwash or Sage Alcohol Free mouthwash, teeth brushing (with Sage Toothette Oral Care, Sodium Bicarbonate Toothpaste and Sage Suction Toothbrush) every 12 hours, deep oral suctioning every 8 hours and prior to oral Endotracheal tube (ET) retaping, and Paroex Oral Rinse chlorohexidine gluconate (15ml) swabbed onto oral surfaces every 12 hours (SICU patients only). Mouth care is documented every two hours.
  Arms: Standard of Care oral care

SUMMARY:
The purpose of this study is to see if a 4 day oral care program in patients who have been on a breathing machine results in better oral health, reduces the amount of certain bacteria in the mouth and reduces infection while in the hospital.

The plan is to test the specific hypotheses that a standardized oral care protocol:

1. Results in improved oral health compared to standard care,
2. Reduces the rate of Staphylococcus aureus / methicillin resistant Staphylococcus aureus, and
3. Reduces the risk of healthcare-associated infections.

DETAILED DESCRIPTION:
Upon meeting inclusion criteria and consenting to participate, the subject will be enrolled in the study. Upon extubation, the subject will be randomly assigned using a computer generated table of random numbers to either the intervention or control group. Daily safety checks including reviewing INR and platelet counts (if performed) will be performed to ensure patient has maintained eligibility for the study.

Study Intervention:

Control Arm:

Current practice in the intensive care units includes the provision of oral care as part of the Ventilator Bundle guideline focused on the reduction of VAP. Currently, the intensive care units utilize a commercially available pre-package oral hygiene kit. This includes mouth care (alcohol free mouthrinse and hydrogen peroxide) with swabs every 2 hours, tooth brushing (suction toothbrush with anti- plaque paste) every 12 hours, deep oral suctioning every 8 hours and prior to ET tube retaping, and chlorohexidine gluconate (15ml) swabbed onto oral surfaces every 12 hours (SICU patients only). Mouth care is documented every two hours.

On the progressive care units and general medical-surgical units, routine oral care is provided as part of the general hygiene care of the units, and based on the clinical determination of the nurse. The selection of oral care techniques currently used on the progressive care units is determined by the level of independence of the patient and oral hygiene needs of the patient. Two techniques are currently being implemented: 1) toothbrushing using a basic toothbrush and basic oral care products provided by the hospital every 12- 24 hours. 2) The prepackaged suctioning kit which includes suction toothbrush with toothpaste and suction oral swabs with alcohol-free mouth rinse, and hydrogen peroxide every 4 hours or based on clinical judgement. Lip moisturizer is applied inside the mouth and on the lips.

Intervention Arm The intervention proposed would include a 4-5 day systematic oral hygiene program provided to patients who are post-extubation. The proposed intervention would begin in the intensive care unit within 24 hours post-extubation and when the patient is determined to be medically stable. The protocol would be initiated with an intensive oral hygiene intervention (see Appendix A) with selected oral hygiene products in the post-extubation period. Following the oral hygiene intervention of the oral cavity, the intervention would continue even if the patient transitions from the intensive care setting to either the progressive care unit or general medical-surgical unit. The intervention will be provided by the Clinical Nurse Specialist (key personnel) from the Division of Critical Care Nursing and Medical-Surgical Nursing. The oral hygiene program will be provided a total of 9 times.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Has required mechanical ventilation for at least 48 hours
* Meets ventilator liberation criteria (PEEP ≤ 8 and FiO2 ≤ 50%)
* Minimum of 3 teeth
* Either the subject or their Legally Authorized Representative is capable of reading, understanding and providing written informed consent.

Exclusion Criteria:

* Non-English speaking
* Allergy to products/components of the oral care protocol
* Oral or maxillofacial surgery, or oral/facial trauma in last three months
* INR > 3.5 or platelet count < 20,000
* Planned hospital discharge within 48 hours
* Current diagnosis of mucositis, or undergoing chemotherapy or radiation therapy
* Presence of Tracheostomy
* Family or physician not in favor of continued medical treatment.
* Unable to give informed consent, and/or lack of availability of an authorized representative who can provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in prevalence of Methicillin-sensitive Staphylococcus aureus (MSSA) in post mechanically ventilated patients as assessed by Oral cultures (Swabs) | Day 1 and 4 days post-extubation
  The overall purpose of this project is to develop an evidence-based oral care protocol for acutely ill hospitalized patients and determine the impact of this protocol on health outcomes in recently extubated patients. The aim is to assess the impact of an oral care protocol on the following rate of oral colonization with Methicillin-sensitive Staphylococcus aureus (MSSA)
Change in prevalence of Methicillin-resistant Staphylococcus aureus (MRSA) in post mechanically ventilated patients as assessed by Oral cultures (Swabs) | Day 1 and 4 days post-extubation
  The overall purpose of this project is to develop an evidence-based oral care protocol for acutely ill hospitalized patients and determine the impact of this protocol on health outcomes in recently extubated patients. The aim is to assess the impact of an oral care protocol on the following rate of MRSA,

SECONDARY OUTCOMES:
Determine infection rate of healthcare acquired infections (MSSA and MRSA) in post mechanically ventilated patients receiving oral care using nasal cultures (Swabs) | 4 days
  Obtain Data on the incidence of new MSSA and MRSA infections in the post-mechanically, ventilated post-ICU patient using nasal cultures (Swabs)
Identify change in patient satisfaction in post mechanically ventilated patients who receive oral care using a Patient satisfaction survey/interview. | 4 days post extubation
  Assess whether there is an increase in patient satisfaction in those receiving the intervention by using Patient satisfaction survey/interview.
Identify change in patient quality of life in post mechanically ventilated patients who receive oral care using the Edmonton Symptom Assessment System quality of life assessment tool. | 4 days post extubation
  Measure change in patient quality of life as reported using the Edmonton Symptom Assessment System quality of life assessment tool of 0 to 10 scale, where 0 represents no symptom and 10 represents the worst possible severity.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Chipps, RN,PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States